CLINICAL TRIAL: NCT00100945
Title: A Phase II Study Of Maintenance ZD1839 (IRESSA) In Patients With Locally Advanced Esophageal Cancer After Treatment Given With Curative Intent
Brief Title: Gefitinib in Treating Patients With Locally Advanced Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0342; NCI-2012-02644 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000407534 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; stage II esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gefitinib (Experimental): Patients receive oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease recurrence or unacceptable toxicity.
  Quality of life is assessed at baseline, 4 weeks, every 12 weeks during study treatment, and then at the end of study treatment.
  Patients are followed every 3 months for up to 5 years.
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well gefitinib works in treating patients with locally advanced esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 1-year overall survival rate in patients with previously treated locally advanced adenocarcinoma of the esophagus or gastroesophageal junction treated with gefitinib as maintenance therapy.

Secondary

* Determine disease-free survival and time to disease recurrence in patients treated with this drug.
* Determine the toxicity of this drug in these patients.
* Determine the quality of life of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease recurrence or unacceptable toxicity.

Quality of life is assessed at baseline, 4 weeks, every 12 weeks during study treatment, and then at the end of study treatment.

Patients are followed every 3 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the esophagus or gastroesophageal junction

  * Locally advanced disease

    * T3 or T4 tumor with no lymph node involvement OR any T stage with local lymph node involvement

      * Celiac node involvement allowed
      * No supraclavicular lymph node involvement
* Received potentially curative chemotherapy, radiotherapy, and/or surgery within the past 1-3 months

  * Patients who received adjuvant chemotherapy or chemoradiotherapy after surgery are eligible provided last treatment was administered within the past 3 months
* No evidence of residual tumor or metastatic disease after undergoing potentially curative therapy

  * No positive margins at the time of prior surgery
  * No measurable or evaluable disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 2.0 mg/dL

Renal

* Creatinine ≤ 2 times upper limit of normal

Cardiovascular

* No New York Heart Association class III or IV heart disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow study drug
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or noninvasive carcinoma

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics

Other

* No prior gefitinib
* No concurrent CYP3A4 inducing agents, including any of the following:

  * Carbamazepine
  * Oxcarbazepine
  * Modafinil
  * Ethosuximide
  * Griseofulvin
  * Nafcillin
  * Phenobarbital
  * Phenylbutazone
  * Phenytoin
  * Primidone
  * Rifampin
  * Hypericum perforatum (St. John's wort)
  * Sulfinpyrazone
* No concurrent antacids 4 hours before or after study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-07; Primary Completion 2007-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
1-year overall survival rate | Up to 12 months

SECONDARY OUTCOMES:
Survival time | Up to 5 years
Disease-free survival | Up to 5 years
Time to disease recurrence | Up to 5 years
Time to treatment failure | Up to 5 years
Quality of life | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (119):
- United States (119):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin

REFERENCES:
- [Derived] Smith RS, Foster NR, Jatoi A, Thome SD, Miller RC. Incidence of Brain Metastasis as First Event in Patients with Esophageal Carcinoma: a Report from Three Prospective Alliance Clinical Trials. J Gastrointest Cancer. 2023 Sep;54(3):846-854. doi: 10.1007/s12029-022-00871-7. Epub 2022 Oct 17. PMID 36251211